CLINICAL TRIAL: NCT00159848
Title: Effectiveness Of An Educational Program To Improve Patients' Satisfaction Regarding Their Management Of Erectile Dysfunction With Sildenafil
Brief Title: Effect Of A Treatment Optimization Program To Improve Satisfaction With Viagra
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: NRA1481115
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction

INTERVENTIONS:
Behavioral: Treatment Optimization Program (educational material)

SUMMARY:
This study will demonstrate if a treatment optimization program has an impact on the satisfaction with Viagra treatment in men with erectile dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Male subjects above age of majority for whom sildenafil is prescribed for the first time within the usual practice of medicine

Exclusion Criteria:

* Male subjects who have used any ED medical treatments over the last month, with the exception of testosterone and/or herbal therapies
* Subjects who do not have the possibility of viewing the video either through a computer, VCR or a DVD

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000
Dates: Start 2003-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Assess the impact of a sildenafil educational program versus usual care on subjects' satisfaction regarding their management of ED with sildenafil as assessed through the validated EDITS questionnnaire after 3 months of treatment

SECONDARY OUTCOMES:
Describe the relationship between the administration of an educational program and the effectiveness of sildenafil; Evaluate the educational program as a tool to help physicians in their management of ED; Estimate the intracluster correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer